CLINICAL TRIAL: NCT02299492
Title: Person-Centered Care Planning and Service Engagement
Acronym: PCCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: University of Pennsylvania (Other); Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PCCP-13-9762
Record Dates: First submitted 2014-11-13; First posted 2014-11-24 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2020-09

CONDITIONS: Severe Mental Illness
Keywords: Mental Health Services
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Person-Centered Care Planning (Experimental): Arm will receive provider level training in Person Centered Care Planning
  Interventions: Other: Person Centered Care Planning
- Treatment as Usual (No Intervention): Arm will receive treatment as usual in community mental health clinic

INTERVENTIONS:
Other: Person Centered Care Planning — PCCP is a manualized provider-based intervention that maximizes consumer choice for adults receiving mental health services. PCCP focuses on engagement and individualized care, thereby enhancing the impact of existing evidence based practices.
  Arms: Person-Centered Care Planning

SUMMARY:
This proposed study addresses the problem of service disengagement within the mental health system. No matter how effective mental health practices are now or become in the future, they are of little value should persons with mental illnesses continue to choose not to receive them. Consumers have attributed their disengagement from care to having poor alliances with care providers, including experiences of not being listened to and not being offered the opportunity to make decisions and collaborate in their own treatment. Person-centered care planning is a field-tested intervention designed to maximize consumer choice and ownership of the treatment process. Providers collaborate with consumers to develop customized plans that identify life goals and potential barriers to achieving them. The proposed study tests the effectiveness of Person-Centered Care Planning (PCCP) designed to target barriers and efficiently implement PCCP throughout an agency. By conducting a randomized controlled trial with 14 community mental health clinics from two states, the study will assess whether PCCP improves service engagement and consumer outcomes. The study will also utilize qualitative methods to understand how care planning impacts service engagement and how implementation processes influence organizational and provider level behavior. Designed to bridge the science to services gap, this study focuses on two priorities identified by the NIMH Diversion of Services and Intervention Research: developing models and methods to implement effective mental health services in the community and the study of personalized mental health care.

DETAILED DESCRIPTION:
Service disengagement is one of the most pervasive and challenging problems currently facing the mental health care system. No matter how effective mental health services are now or become in the future, they are of little value should persons with mental illnesses continue to choose not to receive them. Consumers have attributed their disengagement from care to having poor alliances with care providers, including experiences of not being listened to and not being offered the opportunity to make decisions and collaborate in their own treatment. In response, the mental health system is moving toward a more person-centered model, based upon recovery principles, to engage consumers more actively in their care. While states have embraced this model in theory, they are now looking for guidance as to how best to implement this model in practice, including how to maximize service quality and consumer outcomes given the limited resources available to them for workforce development.

The proposed study tackles this pressing issue by testing the effectiveness of Person-Centered Care Planning (PCCP). By targeting treatment planning - a process that is common across clinical interventions - PCCP has the potential to enhance evidence based practices. PCCP is a field-tested intervention designed to maximize consumer choice and ownership of the treatment process.Providers collaborate with consumers to develop customized plans that identify life goals and potential barriers to achieving them. PCCP is implemented agency-wide through clinical supervisor trainings, which provide an experiential teaching program and tools to translate the practice to frontline clinicians.

Our controlled trial will randomize community mental health centers from two states to receive either PCCP or treatment as usual. The study will conduct surveys of agency providers to assess the impact of PCCP on transformational leadership, recovery orientation, and organizational readiness. Provider PCCP competency associated with the intervention will be measured via provider surveys and client medical record review. Client outcomes will include service engagement, satisfaction with services, adherence, employment, housing, and social support. Client outcomes will be measured using secondary data from agency, state and federal datasets. Qualitative inquiry will be used to better understand the care planning and implementation process associated with the intervention. Focus groups will be conducted with providers and consumers in the experimental sites. The specific aims of the study are:

1. Assess the effectiveness of PCCP. H1: Relative to treatment as usual, a significantly larger proportion of participants receiving PCCP will engage in services, have greater satisfaction with services, and have improved outcomes.
2. Assess the effect of organizational factors on the implementation and effectiveness of PCCP
3. Use qualitative methods to understand how care planning impacts service engagement and how implementation processes influence organizational and provider level behavior.

Designed to bridge the science to services gap, this statewide study focuses on how agencies can bring about the wholesale transformation needed to deliver sustainable person-centered care. This study is the first of its kind to examine the synergy between PCCP, sophisticated organizational change methods, and provider level training, and to document their impact on consumer outcomes. This investigative team brings together experts in PCCP and recovery with experts in services and implementation research to generate valuable guidance for how state systems engaged in the transformation process can best use their limited resources during times of significant fiscal constraint.

ELIGIBILITY:
Inclusion Criteria:

* Receiving services at participating community mental health clinics

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Actual)
Dates: Start 2013-09-01; Primary Completion 2019-02-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Service Engagement | 12 Month
  Consumers attending scheduled appointments at mental health clinics
Service Engagement | 24 Month
  Consumers attending scheduled appointments at mental health clinics

SECONDARY OUTCOMES:
Person Centered Care Competency | 12 Month
  The 32-item Person Centered Care Questionnaire assesses fidelity to the PCCP intervention.
Recovery Orientation | 12 Month
  The Recovery Self Assessment is a 36-item measure assessing the degree to which recovery oriented practices are implemented in an agency.
Person Centered Care Competency | 18 Month
  The 32-item Person Centered Care Questionnaire assesses fidelity to the PCCP intervention.
Recovery Orientation | 18 Month
  The Recovery Self Assessment is a 36-item measure assessing the degree to which recovery oriented practices are implemented in an agency.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Stanhope, PhD, Principal Investigator — New York University
Locations (1):
- New York University, New York, New York, United States

REFERENCES:
- [Derived] Stanhope V, Matthews EB. Delivering person-centered care with an electronic health record. BMC Med Inform Decis Mak. 2019 Aug 22;19(1):168. doi: 10.1186/s12911-019-0897-6. PMID 31438960
- [Derived] Stanhope V, Tondora J, Davidson L, Choy-Brown M, Marcus SC. Person-centered care planning and service engagement: a study protocol for a randomized controlled trial. Trials. 2015 Apr 22;16:180. doi: 10.1186/s13063-015-0715-0. PMID 25897762